CLINICAL TRIAL: NCT00000203
Title: Buprenorphine Maintenance for Opioid Addicts
Brief Title: Buprenorphine Maintenance for Opioid Addicts - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-05626-2; R01DA005626 (NIH); R01-05626-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to evaluate varying doses of buprenorphine for opioid dependence and cocaine abuse.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 1988-08; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Drug use
Withdrawal symptoms
Psychological symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Kosten, M.D., Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, New Haven, Connecticut, United States

REFERENCES:
- [Background] Schottenfeld RS, Pakes J, Ziedonis D, Kosten TR. Buprenorphine: dose-related effects on cocaine and opioid use in cocaine-abusing opioid-dependent humans. Biol Psychiatry. 1993 Jul 1-15;34(1-2):66-74. doi: 10.1016/0006-3223(93)90258-f. PMID 8373940